CLINICAL TRIAL: NCT03915301
Title: VUSCH/PostOperativePainTreatment1
Brief Title: Effective Postoperative Pain Treatment After Sternotomy. Comparison of the Erector Spinae Plane Block vs Conventional Opioid Treatment
Acronym: VUSCH/POPT1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pavol Jozef Safarik University (Other)
Responsible Party: Principal Investigator, Kočan Ladislav, Principal investigator, Pavol Jozef Safarik University
Other Study IDs: 1/2019/VUSCH/EK
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Pain Reliefe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESPB: Erector spinae plane block group
  Interventions: Procedure: Satisfaction assessed by the VAS [followed by its scale information in the Description]
- Opioids: Opioid group
  Interventions: Procedure: Satisfaction assessed by the VAS [followed by its scale information in the Description]

INTERVENTIONS:
Procedure: Satisfaction assessed by the VAS [followed by its scale information in the Description] — Erector spinae plane block provided in thoracic part of spine, VAS scale 0-10

SUMMARY:
Comparison of effect between Erector Spinae plane block and conventional opioid treatment after cardiac surgery

DETAILED DESCRIPTION:
Comparison of effect between Erector Spinae plane block and conventional opioid treatment after cardiac surgery. In group "A" will be erector spinae plane block provided in the thoracic part of the body, under ultrasound control. In the group B will be analgesia provided by Pethidine. Numerical pain score will be recorded every 2 hours, also usage of analgetics will be recorded in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative state after cardiac surgery, Serious pain NRS 8-10

Exclusion Criteria:

* disagreement

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients after cardiac surgery
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-07-20 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with pain treatment assessed by the numerical rating scale VAS | 12 hours
  Pain assessed by VAS 0-10 score

CONTACTS AND LOCATIONS:
Locations (1):
- East Slovak Institute for Cardiovascular Diseases, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided